CLINICAL TRIAL: NCT04218370
Title: LIBERation From AcuTE Dialysis
Acronym: LIBERATE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIBERATED; R01DK122797 (NIH)
Record Dates: First submitted 2019-12-19; First posted 2020-01-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury; Kidney; Disease, Acute; Dialysis Related Complication
MeSH Terms: conditions — Acute Kidney Injury; Disease | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Thrice-weekly intermittent dialysis until pre-specified criteria for recovery are met
  Interventions: Procedure: Dialysis
- Conservative (Experimental): Conservative dialysis strategy--dialysis prescribed only when specific metabolic or clinical indications are met. These indications are: blood urea nitrogen >112 mg/dL (40 mmol/L; blood potassium concentration >6 mmol/L; blood potassium concentration >5.5 mmol/L despite medical treatment; arterial blood gas pH <7.15, or in the absence of an available blood gas, serum bicarbonate <12 mmol/L, acute pulmonary edema due to fluid overload, responsible for hypoxemia requiring oxygen flow rate >5 L/min or equivalent via face mask/tracheostomy mask to maintain SpO2 >95% or requiring FiO2 >50% in patients with tracheostomy already on invasive or non-invasive mechanical ventilation and despite diuretic therapy; clinician judgement
  Interventions: Procedure: Dialysis

INTERVENTIONS:
Procedure: Dialysis — Dialysis treatment, either in the form of hemodialysis or continuous renal replacement therapy (if patient develops hemodynamic instability)

SUMMARY:
The goal of the LIBERATE-D clinical trial is to improve outcomes for patients recovering from dialysis-requiring acute kidney injury (AKI-D). The impact of a conservative dialysis strategy compared to standard clinical practice of thrice-weekly dialysis will be examined to help generate knowledge for how to guide delivery of dialysis to facilitate renal recovery.

DETAILED DESCRIPTION:
Dialysis-requiring acute kidney injury (AKI-D) is a devastating complication among hospitalized patients for which there are no treatments other than supportive care. Recovery of sufficient renal function to stop dialysis is an unequivocally important clinical and patient-oriented outcome. Shortening dialysis duration and increasing the number of AKI-D patients who recover would have a major clinical, public health and cost-saving impact. However, there is currently no evidence to guide the delivery of dialysis to facilitate recovery. The investigators hypothesize that in patients who have AKI-D and who are hemodynamically stable, a conservative dialysis strategy--in which hemodialysis is not continued unless specific metabolic or clinical indications for renal replacement therapy (RRT) are present--will improve the likelihood of renal recovery compared with the current standard clinical practice of thrice-weekly intermittent dialysis. The investigators have conducted a pilot clinical trial to demonstrate the feasibility of this approach. The investigators propose here a 2-center randomized controlled trial to test a conservative dialysis strategy in a larger AKI-D population (N = 220).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Inpatient with AKI-D (intermittent hemodialysis or continuous renal replacement therapy received on at least one calendar day) at least partially due t acute tubular necrosis per the clinical nephrology team
* Hemodynamic stability: not requiring vasopressor support and with planned intermittent dialysis
* Baseline estimated glomerular filtration rate (eGFR) ≥ 15 mL/min/1.73 m2

Exclusion Criteria:

* Nontraditional indication for dialysis (end-stage liver disease awaiting transplantation, fulminant hepatic failure, intoxication)
* Complete nephrectomy as cause of AKI-D
* Kidney transplant during index hospitalization
* Dialysis > 3 months
* Decompensated heart failure requiring left ventricular assist device or continuous inotropic support
* Mechanical ventilation via endotracheal tube
* Hypoxemia requiring significant oxygen support: >5 liters/min via nasal cannula or equivalent via face mask/tracheostomy mask to maintain oxygen saturation > 95%, or requiring fraction of inspired oxygen >50% in patients with tracheostomy requiring invasive or non-invasive ventilation
* Unable to consent and no surrogate decisionmaker available
* Pregnant
* Prisoner
* Clinical team declines to allow study participation
* Anticipated discharge or transfer from study hospital within 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with renal recovery at hospital discharge | Up to 14 days after hospital discharge (to allow for ascertainment of outcome at hospital discharge, which requires a period of sustained dialysis independence)
  Alive and off dialysis at the time of discharge, with sustained independence from dialysis for 14 days. This outcome does not require that all 14 days of sustained independence occur in-hospital.

SECONDARY OUTCOMES:
Number of dialysis sessions/week | Up to 28 days
  Number of dialysis sessions prescribed in each treatment arm, expressed per week.
Dialysis-free days to study day 28 | Up to 28 days
  The number of days that a patient did not need dialysis to study day 28. A patient can only accrue dialysis-free days after the final dialysis session that commences the monitoring period for renal recovery. Subjects who die before study day 28 will be considered to have zero dialysis-free days.

OTHER OUTCOMES:
Renal recovery at day 28 | Up to 42 days (to allow for ascertainment of outcome at day 28, which requires a period of sustained dialysis independence)
  Alive and off dialysis at day 28, with sustained independence from dialysis for 14 days.
Renal recovery | Up to 104 days (to allow for ascertainment of outcome at day 28, which requires a period of sustained dialysis independence)
  Alive and off dialysis at day 90, with sustained independence from dialysis for 14 days.
All-cause in-hospital mortality | Up to date of death from any cause, assessed up to 12 months
  Vital status at the time of hospital discharge
All-cause day 28 mortality | Up to 28 days
  Vital status at day 28 after study enrollment
All-cause day 90 mortality | Up to 90 days
  Vital status at day 90 after study enrollment
Length of hospital stay | Up to date of hospital discharge or death from any cause, whichever comes first, assessed up to 12 months
  Duration of hospital stay after study enrollment
Time to renal recovery | Up to day 90
  Days after study enrollment before renal recovery occurs
Pre-specified adverse events | Up to 28 days
  Adverse events that might be related to the dialysis intervention, including emergent dialysis sessions, intradialytic hypotension and post-dialysis hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Liu, MD, PhD, MAS, Principal Investigator — University of California, San Francisco; Chi-yuan Hsu, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of Califonia, San Francisco, San Francisco, California
  - Washington University in St Louis/Barnes-Jewish Hospital, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu KD, Siew ED, Tuot DS, Vijayan A, Matzumura Umemoto G, Birkelo BC, Lee BJ, Kwong YD, McCoy IE, Delucchi K, Zhuo H, Hsu CY. A Conservative Dialysis Strategy and Kidney Function Recovery in Dialysis-Requiring Acute Kidney Injury: The Liberation From Acute Dialysis (LIBERATE-D) Randomized Clinical Trial. JAMA. 2025 Nov 7:e2521530. doi: 10.1001/jama.2025.21530. Online ahead of print. PMID 41201895
- [Derived] McCoy IE, Liu KD, Ghamarian E, Quenot JP, Zarbock A, Bihorac A, Khoo B, Gallagher MP, Du B, Joannidis M, Kashani K, Tolwani A, Bagshaw SM, Wald R; STandard versus Accelerated initiation of Renal Replacement Therapy in AKI (STARRT-AKI) Investigators. Dialysis Dependence in Standard versus Accelerated Initiation of KRT in AKI: A Post Hoc Analysis. Clin J Am Soc Nephrol. 2025 May 1;20(5):601-607. doi: 10.2215/CJN.0000000672. Epub 2025 Mar 11. PMID 40232884